CLINICAL TRIAL: NCT01352091
Title: A Randomized ,Open Label Study Comparing the Efficacy of Zoladex® Combined With Arimidex® for 3-2 Years After Selective Estrogen Receptor Modulators (SERMs) as an Adjuvant Therapy for 2-3 Years Versus Continuing Tamoxifen up to 5 Years for Premenopausal Early Breast Cancer Patients With Hormone Receptor Positive, Lymph Node Positive or Tumor≥ 4cm.
Brief Title: Adjuvant AI Combined With Zoladex
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Fudan University Shanghai Cancer Center, Fudan University Shanghai Cancer Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CBCSG002
Record Dates: First submitted 2011-05-10; First posted 2011-05-11 (Estimated); Last update posted 2011-05-11 (Estimated); Status verified 2008-04

CONDITIONS: Breast Cancer
Keywords: breast cancer; adjuvant endocrine therapy; AI; Zoladex
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Switch to Zoladex + AI for 3-2 years (Experimental): Patients who took tamoxifen or Fareston for 2-3 years were randomized into 2 groups (335 patients for each group). One group would switch to receive Zoladex 3.6mg depot subcutaneously every month and Aromidex 1mg/d po for another 3-2 years
  Interventions: Drug: Zoladex+AI
- TAM (Experimental): Patients who took tamoxifen or Fareston for 2-3 years were randomized into 2 groups (335 patients for each group). One group would receive TAM 20mg/d treated for 3-2 years.
  Interventions: Drug: TAM

INTERVENTIONS:
Drug: Zoladex+AI — Patients who took tamoxifen or Fareston for 2-3 years were randomized into 2 groups (335 patients for each group). One group would switch to receive Zoladex 3.6mg depot subcutaneously every month and Aromidex 1mg/d po for another 3-2 years
  Arms: Switch to Zoladex + AI for 3-2 years
Drug: TAM — Patients who took tamoxifen or Fareston for 2-3 years were randomized into 2 groups (335 patients for each group). One group would receive TAM 20mg/d treated for 3-2 years.
  Arms: TAM

SUMMARY:
The present study is a randomized open-label -phase III study that aims to compare the efficacy of Zoladex® combined with Aromidex® for 3-2 years after SERMs (tamoxifen and Fareston®) as an adjuvant therapy for 2-3 years with the efficacy of tamoxifen up to 5 years for premenopausal breast cancer women with hormone receptor positive, lymph node positive or tumor ≥4cm. According to St. Gallen's guideline, hormone receptor positive was defined as endocrine responsive and endocrine response uncertain categories (table 3-1), and only those with ER or PR expression undetectable were considered as HR negative. The pathological evaluation of axillary lymph node could be done by sentinel node biopsy (SNB) when axillary nodes were clinically impalpable accompanied with axillary lymph node dissection (ALND) or directly through ALND when axillary nodes appeared to be positive in clinical examination. Based on the operating standard of local medical institution, identifying the numbers of lymph nodes to do the pathological evaluation and to do the dissection of I- or II-station nodes accurately.

ELIGIBILITY:
Inclusion Criteria:

1. All patients must have signed and dated an informed consent form
2. Patients must be female
3. Primary invasive breast cancer pathologically approved by core needle or open biopsy
4. Ipsilateral axillary or internal mammary nodes positive, or tumor size is equal to or larger than 4cm. Definition of nodes positive is according to the staging system of AJCC 6th edition (American Joint Cancer Commission) for breast carcinoma. The micrometastasis must be at least 0.2mm
5. Patients must have undergone standard surgery for primary breast cancer as shown in the following:

   * a standard radical mastectomy or modified mastectomy
   * standard breast conservation surgery (BCS), which is lumpectomy or qaudrantectomy accompany with axillary dissection, and the surgical margins of the resected specimen must be negative. BCS must be followed by standardized adjuvant radiotherapy to the partial conserved breast (delivered after adjuvant chemotherapy completed)
   * Treatment for confirmed breast cancer including the surgery modality listed above, loco-regional radiotherapy after lumpectomy, adjuvant radiotherapy to the chest wall and/or internal mammary nodes and/or supraclavicular lymph nodes, adjuvant chemotherapy
6. adjuvant endocrine therapy of TAM or Fareston must be started within 6 weeks when adjuvant chemotherapy or radiotherapy was finished
7. The date of randomization must be processed after taking TAM or Fareston for 2 or more than 2 years, but not more than 3 years of time
8. Patients taking neo-chemotherapy are eligible, and lymph node status could be identified during surgery before neo-adjuvant chemotherapy or after neo-adjuvant chemotherapy. The definition of lymph node positive is:

   * evaluation of lymph node status before neo-adjuvant chemotherapy must include pathological axillary nodes, internal mammary nodes (pN2b option) or supraclavicular nodes (pN3c option) involved. Micro-metastasis (i.e.≥0.2mm, pN1-pN3c) can be identified by the following method: fine needle aspiration (FNA) or sentinel node biopsy (SNB) or sampling/ total procedure of axillary dissection
   * patients with no nodes positive after neo-adjuvant chemotherapy, lymph node positive must be evaluated during surgery. Its definition was the either of following:

     * According the clinical practice guidelines of the local cancer center, it is acceptable when positive nodes was identified by SNB or axillary dissection
     * There is pathological evidence in lymph nodes positive (pN1-pN3c) during breast surgery after neo-adjuvant chemotherapy
9. Patients diagnosed as occult breast cancer clinically are found to pathologically have primary invasive carcinoma or DCIS with micro-invasive lesion in ipsilateral breast, and primary lesion or axillary node metastasis express ER and/or PR positive
10. Patients with synchronous bilateral cancers are eligible on the condition that If one side is IDC and the other side is DCIS, the IDC side should be of the ER and/or PR positive phenotype and IF two sides are both IDC, they must be ER and/or PR positive phenotype at the same time
11. Hormone receptor positive (≥＋) is defined as detecting ER or PR expression at any time is eligible. The situation of only PR positive and ER negative is eligible, too
12. According to the standard operation principles for clinical practice of local cancer center, patients must be randomized within 4 weeks after definitive physical examination, imaging examination and laboratory testing show no evidence of recurrence or metastasis
13. Based on the study objective, all patients are required to be premenopausal as defined by

    * menstruating actively
    * less than 6 months since last menstrual period (LMP), or patients younger than 40 years of age who became amenorrheic not more than 1 year if the serum free E2、FSH and LH level was premenopausal (according to the reference value of local center).
    * had previous hysterectomy with one or both ovaries left intact are eligible if the serum free E2、FSH and LH level are premenopausal (according to the reference value of local center).
14. patients must have an ECOG performance status of 0 or 1 (0-fully active, able to carry on all pre-disease performance without restriction, 1-restricted in physical strenuous actively but ambulatory)
15. leucocyte count must be ≥3.0*10^9/L and platelet count must be ≥100*10^9/L
16. AST/SGOT or ALT/AGPT must be <3 times the ULN
17. serum creatinine must be <2 times the ULN
18. patients can swallow pills
19. pregnancy testing is negative and are willing to do contraception during the treatment period

Exclusion Criteria:

1. patients with metastatic malignant tumor
2. previous history of asynchronous bilateral breast cancer
3. any previous malignancy in the past 5 years, except for those treated with curative intent, such as carcinoma in situ of the cervix, squamous carcinoma of the skin or basal cell carcinoma of the skin
4. any non-malignant systemic disease which interfere long time follow up
5. history of medical ovarian ablation therapy
6. history of AI therapy
7. severe live dysfunction, Child-Pugh is grade C
8. Occult breast cancer is found pathologically no IDC lesion or only DCIS without micro-invasive lesion in the ipsilateral breast
9. patients with Her-2 overexpression had used, or is using, or intending to use adjuvant trastuzumab
10. severe heart dysfunction, heart functional classification is above Class III Table 2 Child-Pugh score of hepatic cirrhosis

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 670 (Estimated)
Dates: Start 2008-05; Primary Completion 2015-05 (Estimated); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
DFS | 5 Years
  Disease free survival (DFS): DFS related events ware defined as local recurrence, distant metastasis, secondary primary cancer or death, whichever occurred first.during follow up

SECONDARY OUTCOMES:
OS | 5 years
  Overall survival (OS)
Time to distant metastasis | 5 years
  Time to distant metastasis
Bilateral secondary primary breast cancer morbidity | 5 years
  Bilateral secondary primary breast cancer morbidity
DDFS | 5 years
  Distant disease free survival (DDFS)
Osteoporosis related events | 5 years
  Osteoporosis related events ( BMD and bone fracture incidence)
Other adverse events | 5 years
  Other adverse events (Gynecological events, blood lipids, thrombosis, cardiovascular diseases, and etc.)

CONTACTS AND LOCATIONS:
Locations (1):
- FUSCC, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Li JW, Liu GY, Ji YJ, Yan X, Pang D, Jiang ZF, Chen DD, Zhang B, Xu BH, Shao ZM. Switching to anastrozole plus goserelin vs continued tamoxifen for adjuvant therapy of premenopausal early-stage breast cancer: preliminary results from a randomized trial. Cancer Manag Res. 2018 Dec 27;11:299-307. doi: 10.2147/CMAR.S183672. eCollection 2019. PMID 30643455